CLINICAL TRIAL: NCT05489718
Title: A Dose Escalation Phase I Clinical Study to Evaluate the Tolerability and Safety of IBI324 in Subjects With Diabetic Macular Edema(DME)
Brief Title: A Dose Escalation Study of IBI324 in Subjects With Diabetic Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI324A101
Record Dates: First submitted 2022-06-21; First posted 2022-08-05 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treated with different doses of single intravitreal inmection of IBI324 (Experimental)
  Interventions: Biological: IBI324
- treated with different doses of multiple intravitreal inmection of IBI324 (Experimental)
  Interventions: Biological: IBI324

INTERVENTIONS:
Biological: IBI324 — Dose 2 IBI324 of multiple IVT injection
  Arms: treated with different doses of multiple intravitreal inmection of IBI324
Biological: IBI324 — Dose 2 IBI324 of single IVT injection
  Arms: treated with different doses of single intravitreal inmection of IBI324
Biological: IBI324 — Dose 1 IBI324 of single IVT injection
  Arms: treated with different doses of single intravitreal inmection of IBI324
Biological: IBI324 — Dose 3 IBI324 of single IVT injection
  Arms: treated with different doses of single intravitreal inmection of IBI324
Biological: IBI324 — Dose 3 IBI324 of multiple IVT injection
  Arms: treated with different doses of multiple intravitreal inmection of IBI324

SUMMARY:
This study is designed as a Multi-center, open-label, dose escalation phase I trial to evaluate the safety and tolerability of a single and multiple intravitreal injections of IBI324 in subjects with DME

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign informed consent form and comply with visit and study procedures per protocol.
2. Male or female subjects with age of 18~80 yrs.
3. Diagnosis of diabetes mellitus(type 1 or 2), and current regular use of insulin or other injectable drugs or oral anti-hyperglycaemic agent for the treatment of diabetes.
4. Visual impairment was caused by DME involving the macular fovea.
5. Central macular sub-field thickness (CST) ≥320μm according to OCT.
6. BCVA score of 24-73 letters using ETDRS charts (in 4 meters) in the study eye.
7. Female subjects of childbearing age or male subjects with childbearing age female partner agree to take effective contraceptive measures from the screening period to 3 months after the end of treatment.

Exclusion Criteria:

1. Concomitant diseases that may cause subjects fail to respond to the treatment or confuse the interpretation of the study results.
2. PDR in the study eye.
3. Tractional retinal detachment, pre-retinal fibrosis, vitreomacular traction, or epiretinal membrane involving the fovea or disrupting the macular architecture in the study eye.
4. Active rubeosis in the study eye.
5. The equivalent spherical lens≤-8.00D in the study eye.
6. The intraocular pressure>21 mmHg in the study eye.
7. Active ocular or periocular inflammation/infection in either eye.
8. Prior any treatment of following in the study eye:

   * Intravitreal anti-VEGF treatment within 3 months prior to baseline;
   * Intraocular glucocorticoid injection within 3 months prior to baseline;
   * PRP, local/grid laser photocoagulation within 3 months prior to baseline;
   * Any intraocular surgery (e.g. cataract surgery) within 90 days prior to baseline;
   * The eyes were treated with lasik posterior capsulotomy or glaucoma filtration, radiotherapy 30 days before baseline;
9. Currently untreated diabetes mellitus or previously untreated DM subjects who initiated oral or injectable antidiabetic medication or insulin <90 days;
10. HbA1c of >10% within 28 days prior to baseline;
11. Presence of any systemic disease: including but not limited to unstable angina; cerebrovascular accident or transient cerebral ischemia (within 6 months prior to selection); myocardial infarction (within 6 months prior to selection); serious arrhythmia requiring medical treatment; liver, kidney or metabolic diseases; or malignant tumor;
12. History of severe hypersensitivity/allergy to active ingredients or any excipients of the study drug, or fluorescein and povidone iodine;
13. Pregnant or lactating women or women preparing to become pregnant or breastfeeding during the study period;
14. Participated in any clinical study of any other drug within three months prior to enrollment, or attempted to participate in other drug trials during the study;
15. Other conditions unsuitable for enrollment judged by investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Safety evaluation indicators | Through study completion, a maximum of 24 weeks
  Incidence, relatedness and severity of all adverse events, treatment emergent adverse events and serious adverse events b) Changes in central subfield thickness by OCT compared with baseline

SECONDARY OUTCOMES:
The incidence of adverse events | Through study completion, a maximum of 24 weeks
Changes in visual acuity as measured by BCVA compared with baseline | Through study completion, a maximum of 24 week
Changes in the average thickness of the macula in the central 1 mm ETDRS grid (CST) compared with baseline | Through study completion, a maximum of 24 week
Pharmacokinetic (PK) profiles, such as half-life time (t1/2)，etc | Through study completion, a maximum of 24 weeks
  Positive rate of anti-drug antibody
Immunogenicity evaluation indicators | Through study completion, a maximum of 24 weeks
  Positive rate of anti-drug antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang Z, Sun J, Liu K, Tao L, Liu Q, Wu M, Lu S, Deng J, Li L, Qian L, Li X, Sun X. Phase 1 dose-escalation study of IBI324, a VEGF-A/Ang-2 bispecific antibody, for the treatment of diabetic macular oedema. BMJ Open Ophthalmol. 2026 Jan 5;11(1):e002035. doi: 10.1136/bmjophth-2024-002035. PMID 41494748